CLINICAL TRIAL: NCT06193746
Title: Effect of Non-invasive on Lipid Metabolism and Renal Out Comes in Metabolic Syndrome
Brief Title: Laser Efficiency on Metabolic Parameters
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Elbanna, lecturer cardiovascular, Respiratory disorder and geriatric department,, Cairo University
Other Study IDs: P.T.REC/012/004441
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- study group: wear the laser watch on wrist 3times/weak up to 30 minute for 12 weeks ,
  Interventions: Device: non-invasive laser therapy
- control group: taking advises only

INTERVENTIONS:
Device: non-invasive laser therapy — (diode laser, continuous output, in skin contact mode, 0.005W,0.2cm,beam spot area 0.03cm2, 288j/cm ,1800s) in the morning session, we measured lipid profile and kidney function before and after treatment to measure improvement
  Other Names: laser watch
  Groups: study group

SUMMARY:
Non-invasive laser therapy is laser blood irradiation improves many metabolic parameters. So, this study aims to assess the impact of Non-invasive laser therapy on lipid metabolism and renal out comes

DETAILED DESCRIPTION:
The metabolic syndrome is a constellation of interrelated metabolic risk factors especially central obesity, dyslipidemia, hyperglycemia, which all affect worse their kidney function, and all of this causing mortality. This time line requires a quick procedure that will enable us to implement safe and non-invasive therapeutic instruments adjacent therapy for metabolic syndrome cases.

ELIGIBILITY:
Inclusion Criteria:

* The patients have Metabolic syndrome, started more than one year ago.
* BMI ranged 30- 35Kg/m2.
* They are on medical therapy for more than one year.
* Clinically stable.

Exclusion Criteria:

* taking specific drugs uncontrolled diseases
* cardiovascular instability
* sever e autonomic neuropathy
* infection wound,
* burn, allergy or another external injury
* hypothyroidism
* hemorrhagic disorders
* history of cancer
* pregnant women,
* mental illness as schizophrenia or dementia.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the study population selected from out patient of Berket El-haje medical center suffering from metabolic syndrome
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
lipid profile change | 12 weeks following end of treatment
  laboratorial measurement of lipid in one mg/dl of blood
glomerular function range change | 12 weeks following end of treatment
  laboratorial measurement of glomerular function range in one ml of blood/1minute/1.73m2
creatinine change | 12 weeks following end of treatment
  laboratorial measurement of creatinine one mg/DL of blood

CONTACTS AND LOCATIONS:
Locations (1):
- Toka, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No